CLINICAL TRIAL: NCT02835456
Title: Does Micropattern on Urinary Catheter Surface Reduce Urinary Tract Infections?
Acronym: SHARKLET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jahn Ferenc South Pest Teaching Hospital (Other Government)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Principal Investigator, Prof. Peter Tenke, Director, Department of Urology, Jahn Ferenc South Pest Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCSFC028514
Record Dates: First submitted 2016-07-06; First posted 2016-07-18 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Catheter Associated Urinary Tract Infections
Keywords: CAUTI; Biofilm; Urinary tract infections; micropattern; Catheter
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Sharklet Catheter (Active Comparator): Patient requiring indwelling urinary catheter will be randomised into Group A or Group B
  Interventions: Device: Sharklet Catheter insertion
- Group B: Silicone Foley Catheter (Active Comparator): Patient requiring indwelling urinary catheter will be randomised into Group A or Group B
  Interventions: Device: Silicone Foley Catheter insertion

INTERVENTIONS:
Device: Sharklet Catheter insertion
  Arms: Group A: Sharklet Catheter
Device: Silicone Foley Catheter insertion
  Arms: Group B: Silicone Foley Catheter

SUMMARY:
The aim of this study is to determine if the Sharklet catheter, with its unique surface micropattern, reduces infections in participants, when compared to a standard silicone catheter.

DETAILED DESCRIPTION:
The aim of this study is to determine if the Sharklet catheter, with its unique surface micropattern, reduces infections in participants, when compared to a standard silicone catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires a chronic indwelling Foley catheter for at least 3 days.
* Catheters will not remain indwelling greater than 30 days at a time
* Patient is more than 18 years of age
* Patient is able to give informed consent
* Patient is able to attend follow-up sessions

Exclusion Criteria:

* Patient is less than 18 years of age
* Patient is pregnant
* Patient with a known allergy to silicone
* Patient has urinary tract anatomic abnormality that would prevent placement of a standard Foley catheter
* Patient unable to accommodate the catheter
* Patient has an active urinary tract infection (UTI) or other diagnosed infection that is untreated.
* Patient currently taking (or expected to take) more than a single dose of antibiotics for prevention of other infections during the catheter indwell period
* Patient has uncontrolled fecal incontinence (uncontrolled stool/poop passage)
* Patient is unable to feel and/or communicate their symptoms
* Informed consent is unable to be obtained
* Patient is unable or unwilling to comply with the study follow-up schedule
* Patient has a medical condition or disorder that would limit life expectancy to less than 30 days or that may cause non-compliance with the protocol or confound the data analysis
* Any other reason that if in the opinion of the investigator would make the patient unsuitable for enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Catheter scrapings examined for colonization/biofilm burden and compared to the urine screen collected from the participant (cfu/mL) | 12 weeks
  Determine if there will be less adherent bacteria/biofilm to the Sharklet catheter compared to the controls.
Number of symptomatic Urinary tract infections (UTIs) determined by urine culture. | 12 weeks
  Determine number of symptomatic UTIs between the 2 groups as determined by urine culture.

SECONDARY OUTCOMES:
Incidence of bacteremia | 12 weeks
  Incidence of bacteremia following CA-SUTI
Incidence of Crustation | 12 weeks
  Incidence of catheter obstruction/encrustation requiring removal
Incidence of Discomfort | 12 weeks
  Incidence of significant discomfort/pain requiring removal
Surface analysis of the type of bacteria found on each catheter | 12 weeks
  Surface analysis (e.g., Scanning Electron Microscopy) of removed catheters for qualitative assessment of bacterial colonization
Surface analysis of the amount of encrustation | 12 weeks
  Surface analysis (e.g., Scanning Electron Microscopy) of removed catheters for qualitative assessment of encrustation
Surface analysis of the biofilm formation | 12 weeks
  Surface analysis (e.g., Scanning Electron Microscopy) of removed catheters for qualitative assessment of biofilm formation

CONTACTS AND LOCATIONS:
Locations (1):
- Jahn Ferenc South Pest Teaching Hospital, Budapest, Hungary